CLINICAL TRIAL: NCT05505552
Title: Effects of Vitamin K on Lower-extremity Function in Adults With Osteoarthritis: A Randomized Controlled Pilot Trial
Brief Title: Effects of Vitamin K on Lower-extremity Function in Adults With Osteoarthritis:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Tufts Medical Center (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Sarah Booth, Senior Scientist and Center Director, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R21AR080297 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteo Arthritis Knee
Keywords: osteoarthritis; physical function; nutrition
MeSH Terms: conditions — Osteoarthritis | interventions — Vitamin K; Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin K (Experimental): Participants receive 1 mg/d phylloquinone orally for 24 weeks
  Interventions: Dietary Supplement: Vitamin K
- Placebo (Placebo Comparator): Participants receive daily placebo matching phylloquinone for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K — 1 mg/day phylloquinone (vitamin K1)
  Other Names: Phylloquinone
  Arms: Vitamin K
Dietary Supplement: Placebo — Placebo capsule once daily
  Arms: Placebo

SUMMARY:
The overall goal of this pilot randomized trial is to obtain necessary prerequisite data to conduct a randomized controlled intervention to test the effect of vitamin K supplementation on knee osteoarthritis progression and related functional decline. To address critical parameters required to design this larger RCT, we will conduct a double-blind, 2-armed, parallel-group intervention study, with a placebo run-in, in which 50 adults with mild to moderate knee OA and low baseline vitamin K status will be randomly assigned to 1 mg phylloquinone/day or matching placebo, and treated for 6 months. Specifically, we will: (1) compare the effects of 1 mg/day phylloquinone vs. placebo on the non-functional circulating form of MGP; (2) estimate rates of recruitment and retention, follow-up rates and reasons for loss to follow-up, response rates to questionnaires, adherence/compliance rates, and potential for site differences; and (3) determine the responsiveness of the Osteoarthritis Research Society International (OARSI)-recommended performance-based tests of physical function in adults with low vitamin K status and mild to moderate knee osteoarthritis. We will also obtain preliminary data on the distribution of MGP genotype at two clinical sites for effect size generation.

As of February 2025, based on attrition rate below what was initially expected, we revised our planned enrollment from 50 to 35, to achieve the original goal of 30 completers. This was approved by the study sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Male or post-menopausal female (no menses in the last year)
* Plasma phylloquinone <1.0 nmol/L
* Chronic knee discomfort based on affirmative response to the question "During the past 12 months, have you had pain, aching, or stiffness in or around your knee(s) on most days for at least one month?"
* Kellgren-Lawrence (KL) grade 2-3 in at least one knee
* Ability to understand study procedures and to comply with them for the entire length of the study
* Ability to answer questions by phone
* Ability to swallow capsules

Exclusion Criteria:

* KL grade 4 in at least one knee
* Inability to walk
* Cognitive impairment (based on a Montreal Cognitive Assessment Test score ≤ 17)
* Widespread pain
* Malabsorption disorders (e.g. advance liver disease, stage 4 or 5 chronic renal disease, Crohn's disease, celiac sprue)
* Serious medical conditions or impairments that, in the view of the investigator, would obstruct study participation
* Plan to permanently relocate from the greater Boston, MA or Chapel Hill NC areas during the trial period
* Planned knee or hip arthroplasty during the study period
* Undergoing cancer treatment
* < 50 years old
* Circulating phylloquinone ≥ 1.0 nmol/L
* Warfarin (Jantoven) use
* Use of other investigational drugs
* Use of herbal, botanical or vitamin K supplements
* Use of assistive walking devices

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma uncarboxylated matrix gla protein | 24 weeks
  Plasma uncarboxylated matrix gla protein is considered a functional indicator of vitamin K status. We will evaluate how it changes in response to 1 mg/d vitamin K supplementation in adults with low vitamin K status at baseline and with radiographic knee OA.

SECONDARY OUTCOMES:
Plasma phylloquinone | 24 weeks
  Circulating phylloquinone is considered a global indicator of vitamin K status. We will evaluate how it changes in response to 1 mg/d vitamin K supplementation in adults with low vitamin K status at baseline and with radiographic knee OA.

OTHER OUTCOMES:
Lower-extremity function - self reported | 12 and 24 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function index is a disease-specific, self-administered questionnaire, for assessing health status and health outcomes in osteoarthritis of the knee and/or hip. WOMAC function scores range from 0-68, with lower scores reflecting better function.
Lower-extremity function - objective measures | 24 weeks
  40-m fast gait speed, Chair stand test, Stair climb test, Timed-up-and-go test, 6 min walk test are measures of lower-extremity function recommended by the Osteoarthritis Research Society International to test physical performance in people with knee OA.
Knee pain | 12 and 24 weeks
  Knee pain, which is symptomatic of OA, will be evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Measurement of Intermittent and Constant Osteoarthritis Pain (ICOAP) self-reported questionnaires. WOMAC pain scores range from 0-20, with higher scores reflecting more pain. ICOAP scores range from 0-100, with higher scores reflecting more pain.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tufts University, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No